CLINICAL TRIAL: NCT03955367
Title: Pelvic Irradiation Versus Prophylactic Extended-field Irradiation in Selected Patients With Cervical Cancer Treated With Concurrent Chemoradiotherapy: A Multicenter, Open-label, Randomized, Phase 3 Trial
Brief Title: Pelvic RT Versus Prophylactic Extended-field RT in Patients With Cervical Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Peking University First Hospital (Other); Cangzhou Central Hospital (Other); The Second Affiliated Hospital of Dalian Medical University (Other); Gansu Wuwei Tumor Hospital (Other); First Affiliated Hospital of Guangxi Medical University (Other); Harbin Medical University Third Affiliated Hospital (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); First Affiliated Hospital of Chongqing Medical University (Other); Guizhou Provincial People's Hospital (Other); Second Hospital of Jilin University (Other); China-Japan Union Hospital, Jilin University (Other); Jilin Provincial Tumor Hospital (Other); Jiangsu Cancer Institute & Hospital (Other); 940 Hospital of the People's Liberation Army Joint Logistic Support Force (Other); General Hospital of Benxi Iron & Steel Industry Group (Unknown); The Affiliated Hospital of Inner Mongolia Medical University (Other); General Hospital of Ningxia Medical University (Other); Beijing Obstetrics and Gynecology Hospital (Other); Tangshan People's Hospital (Other); Zhongnan Hospital (Other); Second Affiliated Hospital of Xi'an Jiaotong University (Other); First Affiliated Hospital Xi'an Jiaotong University (Other); The Affiliated Tumor Hospital of Xinjiang Medical University (Unknown); Zhejiang Cancer Hospital (Other); The First Affiliated Hospital of Zhengzhou University (Other); Affiliated Cancer Hospital of Zhengzhou University (Unknown); Seventh Medical Center of PLA Army General Hospital (Other); Shengjing Hospital (Other); Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other); Xiangya Hospital of Central South University (Other); Henan Provincial People's Hospital (Other); Xi'an Gaoxin Hospital (Other); West China Second University Hospital (Other); The Forth Affiliated Hospital of Guangxi Medical University (Unknown)
Responsible Party: Principal Investigator, Ke Hu, Vice director of Radiation Oncology Department, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PUMCH-EFI
Record Dates: First submitted 2019-05-11; First posted 2019-05-20 (Actual); Last update posted 2022-02-23 (Actual); Status verified 2022-02

CONDITIONS: Uterine Cervical Neoplasms
Keywords: Uterine Cervical Neoplasms; Extended-field irradiation
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Brachytherapy; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pelvic Irradiation (Active Comparator): Patients receive concurrent chemoradiotherapy. The CTV includes the gross tumor, cervix, uterus, parametrium, upper part of the vagina, and pelvic lymph nodes regions. The upper border of CTV is at the level of aortic bifurcation. A dose of 45-50.4Gy is delivered to CTV with IMRT.
  Interventions: Radiation: Pelvic irradiation; Radiation: Intracavitary brachytherapy; Drug: Concurrent chemotherapy
- Prophylactic EFI (Experimental): Patients receive concurrent chemoradiotherapy. The CTV includes the gross tumor, cervix, uterus, parametrium, upper part of the vagina, pelvic lymph nodes regions and para-aortic lymph nodes region. The upper border of CTV is at the level of renal vessels. A dose of 45-50.4Gy is delivered to CTV with IMRT.
  Interventions: Radiation: Prophylactic extended-field Irradiation; Radiation: Intracavitary brachytherapy; Drug: Concurrent chemotherapy

INTERVENTIONS:
Radiation: Prophylactic extended-field Irradiation — CTV covers pelvis and para-aortic lymph nodes region.
  Other Names: Prophylactic radiotherapy for para-aortic lymph nodes region
  Arms: Prophylactic EFI
Radiation: Pelvic irradiation — CTV covers pelvis.
  Other Names: Pelvic radiotherapy
  Arms: Pelvic Irradiation
Radiation: Intracavitary brachytherapy — The total dose delivered to point A or high-risk CTV is ≥80Gy. For patients with larger-volume cervical tumor, the total dose is ≥85Gy.
  Other Names: Brachytherapy
Drug: Concurrent chemotherapy — Cisplatin based concurrent chemotherapy, including cisplatin as a single agent or cisplatin plus Paclitaxel.
  Other Names: Chemotherapy

SUMMARY:
To investigate the value of prophylactic extended-field irradiation (EFI), we conduct a randomized clinical trial to compare the efficacy and toxicity of pelvic irradiation and prophylactic EFI in selected patients with cervical cancer treated with definitive concurrent chemoradiotherapy. External beam radiation therapy is delivered with intensity-modulated radiation therapy (IMRT).

DETAILED DESCRIPTION:
This is a multicenter, open-label, phase III randomized clinical trial. Cervical cancer patients without evidence of para-aortic metastatic lymph nodes (MLNs) and with at least one of the following characteristics are included in the present study: (a) Number of pelvic MLNs ≥ 2; (b)Short diameter of pelvic MLNs ≥ 1.5cm; (c)Pelvic wall involvement. Patients are randomly assigned to pelvic irradiation group and prophylactic EFI group. Patients in pelvic irradiation group receive pelvic irradiation, intracavitary brachytherapy and concurrent chemotherapy. Patients in prophylactic EFI group receive irradiation for pelvis and para-aortic lymph nodes region, intracavitary brachytherapy and concurrent chemotherapy. The upper border of clinical target volume (CTV) is at the level of renal vessels for patients in prophylactic EFI group. A dose of 45-50.4 Gy is delivered to CTV with IMRT in both groups. Patients receive cisplatin based concurrent chemotherapy (single cisplatin or cisplatin plus paclitaxel). The primary endpoint is progression-free survival.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be informed of the investigational nature of this study and give written informed consent with 30 days before treatment.
2. Age ≥18 years and ≤ 70 years.
3. Patients with newly histologically confirmed cervical cancer, including squamous cell carcinoma, adenocarcinoma and adenosquamous carcinoma, et al.
4. No evidence of para-aortic metastatic lymph nodes (MLNs) on CT, MRI or positron emission tomograph (PET)/CT.*
5. No evidence of distant metastasis (FIGO stage IVB).
6. At least meet one of the following characteristics:

   1. Number of pelvic MLNs ≥ 2;
   2. Short diameter of pelvic MLNs ≥ 1.5cm; *
   3. Parametrial involvement to the pelvic wall ＃.
7. Satisfactory performance: Eastern Cooperative Oncology Group (ECOG) score ≥ 2.
8. Adequate marrow: neutrophile granulocyte count ≥1.5*10^9/L, hemoglobin ≥ 80 g/L, platelet count ≥100*10^9/L.
9. Normal liver and kidney function: Creatinine (Cr) < 1.5 mg/dl, Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST) < 2*upper limit of normal (ULN).

   * MLNs refer to positive lymph nodes confirmed by PET/CT or lymph nodes with short diameter ≥ 1 cm on CT or MRI.

     * Parametrial involvement to the pelvic wall is diagnosed with gynecological examination or MRI;

Exclusion Criteria:

1. With common iliac MLNs.
2. Tumor extended to the lower third of the vagina.
3. Tumor spread to mucosa of the bladder or rectum.
4. Prior surgery (including pelvic or para-aortic lymph nodes resection, except for tumor biopsy), radiotherapy or chemotherapy to primary tumor or nodes.
5. Prior malignancy.
6. History of previous radiotherapy to the abdomen or pelvis.
7. Pregnancy or lactation.
8. Active inflammatory bowel disease, or history of severe stomach or duodenal ulcer.
9. Active infection with fever.
10. Patients with unacceptable risk that intracavitary brachytherapy can not be conducted.
11. Any severe disease which may bring unacceptable risk or affect the compliance of the trial, for example, unstable cardiac disease requiring treatment, renal disease, chronic hepatitis, diabetes with poor control, and emotional disturbance.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 638 (Estimated)
Dates: Start 2019-06-17 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 3-year
  Progression-free survival is defined as the time from randomization to disease progression or death from any cause, whichever is first.

SECONDARY OUTCOMES:
Overall survival | 3-year
  Overall survival is calculated from randomization to death from any cause.
Distant failure-free survival | 3-year
  Distant failure-free survival is defined as the time from randomization to distant metastasis or death from any cause, whichever is first.
Para-aortic lymph nodes failure rate | 3-year
  The incidence of para-aortic lymph nodes failure.
Acute toxicity evaluated with CTCAE 5.0 | From the start of treatment to 3 months after treatment.
  Evaluated with CTCAE 5.0
Late toxicity evaluated with Radiation Therapy Oncology Group (RTOG)/EORTC late radiation morbidity scoring scheme | 3-year
  Evaluated with Radiation Therapy Oncology Group (RTOG)/EORTC late radiation morbidity scoring scheme

CONTACTS AND LOCATIONS:
Overall Officials: Ke Hu, Principal Investigator — Peking Union Medical College Hospital
Locations (2):
- China (2):
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - First Affiliated Hospital Xi'an Jiaotong University, Xi’an, Shanxi

REFERENCES:
- [Background] Wang W, Liu X, Meng Q, Zhang F, Hu K. Prophylactic Extended-Field Irradiation for Patients With Cervical Cancer Treated With Concurrent Chemoradiotherapy: A Propensity-Score Matching Analysis. Int J Gynecol Cancer. 2018 Oct;28(8):1584-1591. doi: 10.1097/IGC.0000000000001344. PMID 30153215